CLINICAL TRIAL: NCT04920864
Title: Using Neuromodulation to Investigate Treatment Pathways Associated With Stress and Substance Use in Opioid Use Disorder
Brief Title: rTMS, Stress and Opioid Use Disorder
Acronym: TOTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor of Psychiatry and Behavioral Neurosciences; and Director, Substance Abuse Research Division, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB-21-01-3111
Record Dates: First submitted 2021-05-30; First posted 2021-06-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: A mixed design study will be used to examine the effects of active rTMS vs. sham (within subject) over one of two locations: 10 Hz dlPFC rTMS (group 1) or 1 Hz mPFC rTMS (group 2) in subjects receiving methadone treatment for OUD. The general rTMS treatment protocol will be the same for both groups and will consist of 2 stimulation sessions per day, separated by ~30min, for 5 days (10 total stimulation sessions per treatment protocol). The sham protocol will be the same except the sham rTMS coil will be used. Participants will be randomly assigned to groups and complete the 2 conditions (active vs. sham rTMS) in random order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham rTMS will consist of inactive figure of 8 coil. The participant, rTMS administrator, and assessors will all be blind to coil type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active 10 Hz dlPFC rTMS (Experimental): 10 Hz dorsolateral prefrontal cortex stimulation for 10 sessions (2 sessions/day X 5 days)
  Interventions: Device: rTMS
- Sham dlPFC rTMS (Sham Comparator): inactive dorsolateral prefrontal cortex stimulation for 10 sessions (2 sessions/day X 5 days)
  Interventions: Device: rTMS
- Active 1 Hz mPFC rTMS (Experimental): 1 Hz medial prefrontal cortex stimulation for 10 sessions (2 sessions/day X 5 days)
  Interventions: Device: rTMS
- Sham mPFC (Sham Comparator): inactive medial prefrontal cortex stimulation for 10 sessions (2 sessions/day X 5 days)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Repetitive transcranial magnetic stimulation

SUMMARY:
Opioid agonist treatments are the gold standard for treating opioid use disorder (OUD). Yet, even effective treatments average only 50% six-month retention. Despite extensive research into treatment options, it remains important to improve understanding of factors that contribute to relapse and identify interventions to mitigate these risks.

Stress-exposure is problematic for people trying to recover from substance use disorders (SUDs) because it weakens inhibition of automatic behaviors and increases drug craving and likelihood of relapse. However, paths through which stress affects behavior are incompletely understood and current SUD treatments do not target effects of stress on drug use.

This project will explore whether repetitive transcranial magnetic stimulation (rTMS) might improve treatment outcomes for people with OUD entering methadone treatment. The investigators will examine the impact of rTMS treatment over one of two theoretically-driven neural targets on substance use and cognitive outcomes associated with treatment success (executive function and emotional arousal).

DETAILED DESCRIPTION:
The Competing Neurobehavioral Decisions Systems (CNDS) model of addiction suggests that people with SUDs have altered function and connectivity in fronto-cortical executive control regions (e.g. dorsolateral prefrontal cortex [dlPFC]) and fronto-cortical limbic control regions (e.g. medial prefrontal cortex [mPFC]). Namely, elevated activity in limbic circuitry results in hypersensitivity to drug cues and stress, and decreased executive control impairs the ability to resist drug urges. The CNDS theoretical framework can guide selection and testing of rTMS targets that could improve understanding of the mechanisms of SUDs and stress-induced drug use. Results from previous research suggest that therapeutic effects of rTMS for SUD could occur via excitation of dlPFC or inhibition of mPFC.

The investigators will administer excitatory (10Hz) dlPFC rTMS and inhibitory (1Hz) mPFC rTMS (through an electromagnetic coil placed against the scalp) coupled with tasks of executive function and emotional arousal during stress and neutral conditions (guided imagery task using personalized scripts) in adults with OUD early in methadone treatment. The investigators will examine and compare how strengthening dlPFC activity or reducing mPFC activity may reverse stress-induced executive and emotional dysfunction, respectively, and improve treatment outcomes in persons with OUD seeking to abstain from opioid use.

A mixed design study will be used to examine the effects of active rTMS vs. sham (within subject) over one of two locations: 10 Hz dlPFC rTMS (group 1) or 1 Hz mPFC rTMS (group 2) in subjects receiving methadone treatment for OUD. The general rTMS treatment protocol will be the same for both groups and will consist of 2 stimulation sessions per day, separated by ~30min, for 5 days (10 total stimulation sessions per treatment protocol). The sham protocol will be the same except the sham rTMS coil will be used. Participants will be randomly assigned to groups and complete the 2 conditions (active vs. sham rTMS) in random order. Immediately prior to and after each 5-day rTMS treatment protocol, participants will attend an assessment visit when they will complete multiple tasks during both stress (guided imagery stressor) and neutral conditions. These tasks are designed to measure executive function, emotional arousal, and drug-seeking behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-5 criteria for OUD;
2. In methadone or buprenorphine treatment
3. Age 21-70 yr;
4. Right handed;
5. Males and non-pregnant/non-lactating females;
6. Cognitively intact (total IQ score >80);
7. Use alcohol and/or marijuana <4 times per week; each "time" should consist of <2 marijuana "joint" equivalent and <4 alcoholic drinks.

Exclusion Criteria:

1. Acutely under the influence of any substance (except methadone or buprenorphine) during session;
2. Current, regular (>2 times/week) use of illicit drugs other than opioids (except cannabis);
3. Any past 24 hour use of drugs other than opioids or nicotine;
4. Urinalysis positive for pregnancy;
5. Medical conditions prohibiting use of rTMS;
6. Lifetime psychotic, bipolar, or potentially antisocial personality disorder;
7. Untreated or uncontrolled past-year diagnosis of major depression, generalized anxiety disorder, obsessive compulsive disorder, or post traumatic stress disorder;
8. Past-month SUD other than OUD or tobacco use disorder;
9. Acute/unstable illness making it unsafe for participation;
10. Any prohibited medications including: medications that lower seizure threshold, certain psychiatric medications, or prescription pain medications;
11. Chronic head or neck pain;
12. Past-month participation in a research study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wisconsin Card Sorting Task perseverance score | change from pre-intervention (day 0) to post-intervention (day 5) in the sham and active conditions
  Wisconsin Card Sorting Task perseverance measures cognitive flexibility as an index of executive function. Higher scores reflect better outcome.
Emotional Arousal task rating | change from pre-intervention (day 0) to post-intervention (day 5) in the sham and active conditions
  Average unpleasantness and arousal ratings in response to aversive pictures from the International Affective Picture System (IAPS). Lower unpleasantness and arousal scores reflect better outcome.
Opioid progressive ratio breakpoint | change from pre-intervention (day 0) to post-intervention (day 5) in the sham and active conditions
  Opioid ($10 unit dose) vs. money ($2) hypothetical 10-trial choice task progressive ratio breakpoint is the highest response requirement completed for the drug on an exponentially increasing schedule of reinforcement, where the subject has to click the mouse an increasing number of times to earn drug or money. Lower breakpoint scores reflect better outcome.
Treatment success | change from sham to active condition (randomized to occur on days 6-12 and 18-24, respectively)
  Number of days of opioid use (based on timeline followback interview) during the 7 days following each 5-day rTMS (active and sham) period. Fewer days of opioid use reflect better outcome.

SECONDARY OUTCOMES:
Digit Span total score | change from pre-intervention (day 0) to post-intervention (day 5) in the sham and active conditions
  Digit Span (forward and backward) measures the extent of verbal working memory as an index of executive function. Higher scores reflect better outcome.
Monetary delay discounting | change from pre-intervention (day 0) to post-intervention (day 5) in the sham and active conditions
  Brief version of delay discounting task measures the immediate vs. delayed value of money. Higher area-under-the-curve scores (preference for delayed money) reflect better outcome.
State-Trait Anxiety Inventory state anxiety total score | change from pre-intervention (day 0) to post-intervention (day 5) in the sham and active conditions
  State anxiety subscale score of the State-Trait Anxiety Inventory. Lower scores reflect better outcome.
Positive and Negative Affect Scale total score | change from pre-intervention (day 0) to post-intervention (day 5) in the sham and active conditions
  Positive and Negative Affect Scale measures both positive and negative affect. Lower total negative affect scores reflect better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Greenwald, PhD, Study Director — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No